CLINICAL TRIAL: NCT02063178
Title: Dissemination of the Look Ahead Weight Management Treatment in the Military
Acronym: FITBLUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); United States Air Force (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK097158-01 (NIH); 1R01DK097158-01 (NIH)
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-09

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counselor-Initiated (Experimental): Participants will receive 28 telephone sessions over a 12 month period by interventionists trained in behavior change skills and motivational interviewing techniques. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be encouraged to replace 2 meals and a snack with meal replacements (provided). Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week. The Toolbox includes additional treatment options (e.g., food scales, exercise videos, cookbooks) for those who wish to take advantage of them. There will be several challenges that will provide a specific goal (e.g. increase self-monitoring), with a small award for completion.
  Interventions: Behavioral: Phone-based sessions (28 total) on a structured schedule; Behavioral: Weight self-monitoring; Behavioral: Dietary and physical activity self-monitoring; Behavioral: Scheduled tailored interventionist feedback; Behavioral: Dietary goals; Behavioral: Meal replacements; Behavioral: Physical activity goals; Behavioral: Toolbox; Behavioral: Challenges
- Self-Paced (Active Comparator): The Self-paced group uses a less intense approach, where the participants can receive the same telephone counseling sessions as the counselor-initiated group, only if they call the counselor. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail only upon request. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week.
  Interventions: Behavioral: Phone-based sessions upon request; Behavioral: Weight self-monitoring; Behavioral: Dietary and physical activity self-monitoring; Behavioral: Dietary goals; Behavioral: Physical activity goals; Behavioral: Tailored interventionist feedback upon request

INTERVENTIONS:
Behavioral: Phone-based sessions (28 total) on a structured schedule — 28 sessions will be reviewed weekly and then bi-weekly with a trained motivational interviewing counselor for those individuals randomly assigned to the counselor-initiated condition.
  Arms: Counselor-Initiated
Behavioral: Phone-based sessions upon request — For those individuals randomly assigned to the self-paced condition, the 28 sessions are still available to them, the participant has to call to initiate sessions.
  Arms: Self-Paced
Behavioral: Weight self-monitoring — Each randomized participant will be given a Body Trace scale that will electronically record their weight.
Behavioral: Dietary and physical activity self-monitoring — Each randomized participant will be given a free account to Lose It! Premium, an online food/activity diary for self-monitoring.
Behavioral: Scheduled tailored interventionist feedback — Randomly assigned participants to the counselor-initiated condition will receive feedback on their progress throughout their sessions with their assigned interventionist.
  Arms: Counselor-Initiated
Behavioral: Dietary goals — Each randomized participant will receive a daily calorie goal range based on their current weight, gender, and BMI.
Behavioral: Meal replacements — Randomized participants will receive coupons for meal replacements including oatmeal and popcorn.
  Arms: Counselor-Initiated
Behavioral: Physical activity goals — Each participant will complete the Global Physical Activity Questionnaire which will determine their weekly exercise goals.
Behavioral: Toolbox — The toolbox includes additional treatment options for those who wish to take advantage of them. Items may include: food scales, cookbooks, etc. These items may be checked out and must be returned prior to the completion of the study.
  Arms: Counselor-Initiated
Behavioral: Challenges — There will be several challenges designed to increase participant interest and provide a specific goal (e.g., increase self-monitoring). Participants who successfully completed the challenges will be given a small award.
  Arms: Counselor-Initiated
Behavioral: Tailored interventionist feedback upon request — Randomly assigned participants to the self-paced condition have the option to receive feedback on their progress upon request.
  Arms: Self-Paced

SUMMARY:
Purpose: This study aims to take the procedural and research-based lessons learned from a pilot weight loss intervention (IRB # 13-02563-XP), conducted by The University of Tennessee Health Science Center in 2013, and apply them to the current study of 204 active duty military personnel. The pilot study translated and tailored the Look Ahead weight loss intervention to an overweight/obese active duty U.S. Air Force population, while accommodating the lifestyle and environment that is unique to military members and evaluate materials and procedures used.

Rationale: Being overweight is now by far the leading medical reason for rejection in the military. Unfortunately, the impact of weight problems on the military does not stop with those turned away from military service. From 1998 to 2008, the Armed Forces Health Surveillance Center reported the percent of active military members who experienced medical encounters for overweight or obesity significantly increased. The estimated total days of work lost from absenteeism associated with active-duty personnel who are overweight or obese was 658,000. Using Department of Defense (DOD) estimates of average daily based, it was estimated that overweight and obesity costs the DOD $103 million dollars in health care costs annually. Note this estimate is for active duty personnel only. Furthermore, obesity is a major cause for the discharge of uniformed personnel.

The current study is inspired by the successful Look Ahead trial, a behavioral science obesity intervention treatment program that included: a collaborative approach, education, behavioral support, and motivational interviewing. The unique nature of this weight reduction study is significant. To our knowledge, there had not been a successful translation of a highly efficacious obesity treatment in the military until The University of Tennessee Health Science Center implemented a pilot version of the Fit Blue program for active duty U.S. Air Force members in 2013. Following a successful pilot and extant results from the Look Ahead trial, Investigators expect success during the full scale Fit Blue study.

DETAILED DESCRIPTION:
This study is a weight loss intervention program tailored to a military population. Investigators will randomize 204 consented participants to either an intensive counselor-initiated weight loss intervention or a self-paced weight loss intervention. Neither of the aforementioned conditions are controls and both treatments are expected to result in weight reduction.

Procedures: This is a two-arm individually randomized trial. The Counselor-initiated group will follow a more intense counselor-initiated approach, where the counselor schedules weekly telephone sessions and contacts them directly. The Self-paced group uses a less intense approach, where the participants can receive the same telephone counseling sessions as the counselor-initiated group, only if they call the counselor.

Potential participants will be recruited through the use of advertisements, electronic bulletins, emails, newspapers, and word-of-mouth. Prior to randomization, interested individuals will complete a phone screening, informed consent, two in-person data collection visits and obtain medical clearance, as well as participate in 1 week of dietary and physical activity self-monitoring.

The randomized participants will spend the next year involved in study interventions (either the Counselor-Initiated intervention or the Self-Paced intervention), diet and exercise self-monitoring, daily weighing, and may also include telephone counseling sessions.

The follow-up data collection visits will occur at 4 and 12 months after randomization. At these visits, physical measurements will be collected (i.e. height, weight, abdominal circumference, blood pressure and heart rate) and participants will complete various questionnaires. A Quality of Life questionnaire will also be administered by study personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military personnel at Joint Base San Antonio in the San Antonio, Texas area
2. BMI > 25kg/m2
3. English speaking
4. Clearance by healthcare provider for participation in study
5. >18 years of age
6. Participants have at least one year left on their duty assignment at enrollment

Exclusion Criteria:

1. No access to a computer for self-monitoring in Lose It! or email feedback from counselor
2. Scheduled extended leave away from the San Antonio area in the next 13 months (i.e. planned Permanent Change of Station/Temporary Duty Assignment/deployment)
3. More than one failure of military-proctored physical fitness test on the last 12 months
4. Uncontrolled hypertension defined as Blood pressure > 140/90
5. A member of the same household is already a FitBlue participant
6. Disability or condition that would limit physical activity
7. Current use of a weight loss medication
8. History of significant kidney or liver disease
9. History of uncontrolled thyroid disease or pheochromocytoma
10. Malignancy in last 5 years
11. History of diabetes treated with a medication that could cause hypoglycemia
12. Pregnancy, child birth within the last 6 months, breastfeeding for less than 6 months postpartum, or planning to become pregnant during the study follow-up time (12 months)
13. Presence of an unstable psychiatric condition
14. Severe asthma, bronchitis, or emphysema that precludes exercise
15. History of bariatric surgery or history of significant recent weight loss ( > 10 pounds in past 3 months)
16. Other medical or behavioral factors that in the judgement of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
17. History of cerebral, coronary, or peripheral vascular disease, uncontrolled cardiac arrhythmia, or uncontrolled congestive heart failure in past 12 months
18. Lack of access to telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Krukowski, PhD, Principal Investigator — University of Tennessee
Locations (1):
- Wilford Hall Ambulatory Surgical Center/Lackland Air Force Base, San Antonio, Texas, United States

REFERENCES:
- [Derived] Farage G, Simmons C, Kocak M, Klesges RC, Talcott GW, Richey P, Hare M, Johnson KC, Sen S, Krukowski R. Assessing the Contribution of Self-Monitoring Through a Commercial Weight Loss App: Mediation and Predictive Modeling Study. JMIR Mhealth Uhealth. 2021 Jul 14;9(7):e18741. doi: 10.2196/18741. PMID 34259635
- [Derived] Fahey MC, Klesges RC, Kocak M, Gladney LA, Talcott GW, Krukowski RA. Counselor Efficiency at Providing Feedback in a Technology-Based Behavioral Weight Loss Intervention: Longitudinal Analysis. JMIR Form Res. 2021 May 5;5(5):e23974. doi: 10.2196/23974. PMID 33949954
- [Derived] Manz KC, Waters TM, Clifton HE, Kocak M, Klesges RC, Talcott GW, Krukowski RA. Cost-Effectiveness of a Weight Loss Intervention: An Adaptation of the Look AHEAD Lifestyle Intervention in the US Military. Obesity (Silver Spring). 2020 Jan;28(1):89-96. doi: 10.1002/oby.22681. Epub 2019 Nov 26. PMID 31773873
- [Derived] Pebley K, Klesges RC, Talcott GW, Kocak M, Krukowski RA. Measurement Equivalence of E-Scale and In-Person Clinic Weights. Obesity (Silver Spring). 2019 Jul;27(7):1107-1114. doi: 10.1002/oby.22512. Epub 2019 Jun 5. PMID 31168928
- [Derived] Fahey MC, Klesges RC, Kocak M, Wayne Talcott G, Krukowski RA. Changes in the Perceptions of Self-weighing Across Time in a Behavioral Weight Loss Intervention. Obesity (Silver Spring). 2018 Oct;26(10):1566-1575. doi: 10.1002/oby.22275. PMID 30277031
- [Derived] Krukowski RA, Hare ME, Talcott GW, Gladney LA, Johnson KC, Richey PA, Kocak M, Keller PL, Hryshko-Mullen A, Klesges RC. Dissemination of the Look AHEAD Intensive Lifestyle Intervention in the United States Military: A Randomized Controlled Trial. Obesity (Silver Spring). 2018 Oct;26(10):1558-1565. doi: 10.1002/oby.22293. PMID 30277030
- [Derived] Fahey MC, Hare ME, Talcott GW, Kocak M, Hryshko-Mullen A, Klesges RC, Krukowski RA. Characteristics Associated With Participation in a Behavioral Weight Loss Randomized Control Trial in the U.S. Military. Mil Med. 2019 Mar 1;184(3-4):e120-e126. doi: 10.1093/milmed/usy199. PMID 30125001
- [Derived] Krukowski RA, Hare ME, Talcott GW, Johnson KC, Richey PA, Kocak M, Balderas J, Colvin L, Keller PL, Waters TM, Klesges RC. Dissemination of the Look AHEAD intensive lifestyle intervention in the United States Air Force: study rationale, design and methods. Contemp Clin Trials. 2015 Jan;40:232-9. doi: 10.1016/j.cct.2014.12.014. Epub 2014 Dec 26. PMID 25545025

RESULTS

PARTICIPANT FLOW:
Groups:
- Counselor-Initiated: Will receive 28 telephone sessions over a 12 month period by interventionists trained in behavior change skills and motivational interviewing techniques. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be encouraged to replace 2 meals and a snack with meal replacements (provided). Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week. The Toolbox includes additional treatment options (e.g., food scales, exercise videos, cookbooks) for those who wish to take advantage of them. There will be several challenges that will provide a specific goal (e.g. increase self-monitoring), with a small award for completion.
- Self-Paced: Uses a less intense approach, where the participants can receive the same telephone counseling sessions as the counselor-initiated group, only if they call the counselor. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail only upon request. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week.
Period: Overall Study
Arm/Group | Counselor-Initiated | Self-Paced
Started | 124 | 124
Completed | 95 | 77
Not Completed | 29 | 47

BASELINE CHARACTERISTICS:
Groups:
- Counselor-Initiated: Will receive 28 telephone sessions over a 12 month period by interventionists trained in behavior change skills and motivational interviewing techniques. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be encouraged to replace 2 meals and a snack with meal replacements (provided). Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week. The Toolbox includes additional treatment options (e.g., food scales, exercise videos, cookbooks) for those who wish to take advantage of them. There will be several challenges that will provide a specific goal (e.g. increase self-monitoring), with a small award for completion.
  Phone-based sessions (28 total) on a struct
- Total: Total of all reporting groups
Arm/Group | Counselor-Initiated | Self-Paced | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 124 | 124 | 248
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (8.2) | 33.8 (6.8) | 34.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 63 | 63 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 31 | 56
  Not Hispanic or Latino | 99 | 93 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 26 | 23 | 49
  Caucasian | 79 | 84 | 163
  Other | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 124 | 124 | 248
Weight [Mean (Standard Deviation); unit: kg] — Measured weight on a calibrated scale
  kg | 88.0 (12.9) | 90.0 (15.5) | 89.0 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Loss (Baseline to 12 Months)
Description: The primary data analysis will adhere to the intention-to-treat principle and in the final analysis, the participants will be categorized according to their initial randomization. Investigators will be using the baseline weight as a covariate in the final primary model where the two arms will be compared in terms of the percentage of weight loss.
Time Frame: 12 month intervention
Measure: Mean (Standard Deviation); unit: percent weight loss
Arm/Group | Counselor-Initiated | Self-Paced
Number analyzed (Participants) | 124 | 124
percent weight loss | 2.1 (4.7) | 0.0 (4.0)
Statistical Analysis 1: Comparison: Counselor-Initiated vs Self-Paced; This randomized clinical trial was designed to have 90% power to detect a 4% weight loss percent difference at 12 months between the two study arms; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.1

2. Secondary Outcome: The Relationship Between Attendance and Percent Weight Loss
Description: Evaluating the impact of intervention session attendance on percent weight loss outcome, as a measure of adherence.
Time Frame: 12 month intervention
Measure: Number; unit: spearman rho correlation
Groups:
- Counselor-Initiated: 28 telephone sessions over a 12 month period by interventionists trained in behavior change skills and motivational interviewing techniques. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be encouraged to replace 2 meals and a snack with meal replacements (provided). Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week. The Toolbox includes additional treatment options (e.g., food scales, exercise videos, cookbooks) for those who wish to take advantage of them. There will be several challenges that will provide a specific goal (e.g. increase self-monitoring), with a small award for completion.
  Phone-based sessions (28 total) on a structured schedule
- Self-Paced: Participants can receive the same telephone counseling sessions as the counselor-initiated group, only if they call the counselor. Participants will be asked to monitor food intake and physical activity using the LoseIt website/app and weight daily using a Body Trace e-scale. Participants will receive feedback on self-monitoring through e-mail only upon request. Dietary goals will be based on weight and participants' weight-loss progress. Participants will be asked to gradually increase their moderate to vigorous exercise to 225-250 minutes per week.
  Phone-based sessions upon request: For those individuals randomly assigned to the self-paced condition, the 28 sessions are still available to them, the participant has to call to initiate sessions.
  Weight self-monitoring: Each randomized participant will be given a Body Trace scale that will electronically record their weight.
  Dietary and physical activity self-monitoring: Each randomized p
Arm/Group | Counselor-Initiated | Self-Paced
Number analyzed (Participants) | 124 | 124
spearman rho correlation | 0.49 | -0.10
Statistical Analysis 1: Comparison: Counselor-Initiated vs Self-Paced; The association between weight change percent and attendance was described using Spearman rank correlation; Test type: Other — Correlation; p < 0.0001, Correlation

3. Secondary Outcome: The Relationship Between Dietary and Physical Activity Self-monitoring Adherence and Percent Weight Loss
Description: We will evaluate the impact of dietary and physical activity self-monitoring adherence (using Lose It website/app) on weight loss outcome.
Time Frame: 12 month intervention
Measure: Number; unit: Spearman's rho correlation
Groups:
- Counselor-Initiated: * 28 telephone sessions over a 12 month period by interventionists trained in behavior change skills and motivational interviewing techniques
  * Monitor food intake and physical activity using the LoseIt website/app and weigh daily using a Body Trace e-scale
  * Feedback on self-monitoring through e-mail.
  * Dietary goals will be based on weight and participants' weight-loss progress.
  * Encouraged to replace 2 meals and a snack with meal replacements (provided).
  * Gradually increase moderate to vigorous exercise to 225-250 minutes per week.
  * Toolbox with additional treatment options (e.g., food scales, exercise videos, cookbooks)
  * Challenges that will provide a specific goal (e.g. increase self-monitoring), with a small award for completion.
Arm/Group | Counselor-Initiated | Self-Paced
Number analyzed (Participants) | 124 | 124
Spearman's rho correlation | 0.41 | 0.05
Statistical Analysis 1: Comparison: Counselor-Initiated; Test type: Other; p < 0.0001, Correlation

4. Secondary Outcome: The Relationship Between Self-weighing on Weight Loss
Description: We will also evaluated the impact of self-weighing (using Body Trace e-scales) on weight loss outcomes.
Time Frame: 12 month intervention
Measure: Number; unit: spearman's rho correlation
Arm/Group | Counselor-Initiated | Self-Paced
Number analyzed (Participants) | 124 | 124
spearman's rho correlation | 0.41 | -0.11
Statistical Analysis 1: Comparison: Counselor-Initiated; Test type: Other; p < 0.0001, Correlation

ADVERSE EVENTS:
Time Frame: 13 months
Description: Participants were asked about adverse events at every data collection visit and if during an intervention session they mentioned a potential adverse event, the interventionist gathered details.
Arm/Group | Counselor-Initiated | Self-Paced
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 5/124 | 5/124
Other Adverse Events (participants affected / at risk) | 75/124 | 55/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Counselor-Initiated (N=124) | Self-Paced (N=124)
Gastric Carcinoid Tumor (Gastrointestinal disorders) | 1 (1) | 0 (0)
Third degree burns (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Kidney problems secondary to antibiotics and dehydration while being treated for an ear infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubal ligation (Surgical and medical procedures) | 0 (0) | 1 (1)
New diagnosis of prostate cancer with prostatectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) — After running, investigation did not find a cause
Tibial osteotomy and osteochondral allograft transfer (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Counselor-Initiated (N=124) | Self-Paced (N=124)
Ankle injury (Musculoskeletal and connective tissue disorders) | 13 (13) | 9 (9)
Back injury (Musculoskeletal and connective tissue disorders) | 17 (17) | 17 (17)
Common cold (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 6 (6)
Foot injury (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (10)
Knee injury (Musculoskeletal and connective tissue disorders) | 13 (14) | 12 (12)
Wrist injury (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT02063178/Prot_SAP_000.pdf